CLINICAL TRIAL: NCT03452670
Title: Contemplative Well-being Apps for the Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jennifer Mascaro, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00088349
Record Dates: First submitted 2018-02-13; First posted 2018-03-02 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Social Behavior; Depression; Inflammation
Keywords: Workplace; Applications; Anxiety; Burnout; Meditation; Mindfulness
MeSH Terms: conditions — Social Behavior; Depression; Inflammation; Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The waitlist group will be maintained as a control group throughout all assessments and will be provided enrollment in the mindfulness app at the end of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be blinded by study ID# during data collection and management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Participants in this group will use a contemplative wellness application for 8 weeks.
  Interventions: Behavioral: Active Group
- Waitlist Group (Other): The waitlist group will receive no intervention during the study but will be able to use the wellness application after completion of the study.
  Interventions: Other: Waitlist Group

INTERVENTIONS:
Behavioral: Active Group — Participants will be provided with a contemplative well-being application (CWA) which will facilitate meditation for 10 minutes daily during the 8 week study period.
  Arms: Active Group
Other: Waitlist Group — The waitlist group will be maintained as a control group throughout all assessments and will be provided enrollment in CWA at the end of the 8 week study period.
  Arms: Waitlist Group

SUMMARY:
The study will examine the use and impact of a meditation app delivered to adult workforce populations facing extreme time demands. Enrollees will be randomized to either app or a wait-list group, and will be assessed in terms of job and daily functioning, well-being, and biomarkers of immune function and stress physiology, and neural structure and function prior to randomization and again at multiple time points after participants commence app engagement. In order to assess efficacy, we will examine the longitudinal changes in all measures in both the mindfulness group, compared to wait-list control group.

DETAILED DESCRIPTION:
Over the last 25 years, research on contemplative practices, a family of practices including mindfulness meditation and yoga, has advanced in domains both clinical and basic, motivated by burgeoning evidence of their efficacy for remediating psychopathology and augmenting well-being and resilience. However, much of this research has examined the effects of scheduled group interventions, delivered in-person by instructors over the course of several weeks. Far less research has looked at the delivery method that is most common and arguably most sustainable for busy adults, namely, smart phone delivered Contemplative Applications (apps) for Well-being (CWAs). The proposed study will examine the use and impact of an app delivered to populations facing extreme time demands.

ELIGIBILITY:
Inclusion Criteria:

* Emory Healthcare and University employees, Cox Enterprises employees, and Emory students

Exclusion Criteria:

* For students and employees in the biomarker sub-study, participants will be studied only if they pass the Society of Magnetic Resonance Imaging standardized MRI screening protocol (exclusions for ferrous metal in any part of body, such as pacemakers, cochlear implants, surgical clips or metal fragments, serious medical conditions, claustrophobia)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Change in Incivility in Nursing Education Revised Survey score | Baseline, Week 8
  The Incivility in Nursing Education Revised Survey contains 24-items asking students about behaviors they exhibited or witnessed in the past 12 months (for example, "Students made rude gestures or nonverbal behaviors towards others"). Respondents indicate how often these behaviors occurred by selecting from 1 = Never, 2 = Rarely (only once or twice), 3 = Sometimes (approximately once per month), or 4 = Often (more than once per month). Total scores can range from 24 to 96, with higher scores indicating more incivility performed or witnessed.

SECONDARY OUTCOMES:
Change in School-Burnout Inventory score | Baseline, Week 8
  The School-Burnout Inventory is a 9-item survey asking students about how much burnout they have felt in the past month (for example, "I feel overwhelmed by my schoolwork"). Respondents indicate the degree to which they agree with each statement on a scale of 1 to 6 where 1 = completely disagree and 6 = completely agree. Total scores can range from 9 to 54, with higher scores indicating more burnout.
Change in Depression score on the Depression Anxiety and Stress Scale (DASS) | Baseline, Week 8
  The Depression Anxiety and Stress Scale (DASS) is a 42-item survey asking about feelings of depression and anxiety that the respondent has experienced in the past week (for example, "I found myself getting upset at quite trivial things"). Respondents indicate the degree to which they agree with each statement on a scale of 0 to 3 where 0 = does not apply to me at all and 3 = applied to me very much, or most of the time. The depression subscale includes 14 items. A score of 0-9 indicates no depression, 10-13 indicates moderate depression, 14-20 is moderate depression, 21-27 is severe depression and scores of 28 and above indicate extremely severe depression.
Change in Anxiety score on the Depression Anxiety and Stress Scale (DASS) | Baseline, Week 8
  The Depression Anxiety and Stress Scale (DASS) is a 42-item survey asking about feelings of depression and anxiety that the respondent has experienced in the past week. Respondents indicate the degree to which they agree with each statement on a scale of 0 to 3 where 0 = does not apply to me at all and 3 = applied to me very much, or most of the time. The depression subscale includes 14 items. A score of 0-7 indicates no anxiety, 8-9 indicates moderate anxiety, 10-14 is moderate anxiety, 15-19 is severe anxiety and scores of 20 and above indicate extremely severe anxiety.
Change in Empathic Accuracy (EA) Task | Baseline, Week 8
  The Empathic Accuracy (EA) Task is a dynamic video assessment that asks participants to continuously rate the emotions of others as they tell emotional autobiographical stories. Empathic accuracy is the correlation between feelings of the story-tellers in the video and what the participants perceive the story-tellers feelings to be.
Change in gray matter density in the brain stem | Baseline, Week 8
  The researchers will acquire a high-resolution T1-weighted MRI scan of the whole brain and brain stem from vertex to approximately 2.5 cm below the lower rim of the cerebellum. Gray matter density in the brain stem, with particular focus on the dorsal motor nucleus of vagus nerve and the nucleus of the solitary tract will be measured.
Change in white matter density in the brain stem | Baseline, Week 8
  The researchers will acquire a high-resolution T1-weighted MRI scan of the whole brain and brain stem from vertex to approximately 2.5 cm below the lower rim of the cerebellum. White matter density in the brain stem, with particular focus on the dorsal motor nucleus of vagus nerve and the nucleus of the solitary tract will be measured.
Change in Gene (mRNA) expression in peripheral blood mononuclear cells (PBMCs) | Baseline, Week 8
  Gene (mRNA) expression in PBMCs, focusing on a profile of genes with known involvement in immune function, will be analyzed using the Illumina Human HT-12 BeadArrays.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mascaro, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Wesley Woods Health Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No